CLINICAL TRIAL: NCT03422185
Title: Understanding Local Determinants of Cardiovascular Disease and Diabetes to Inform Novel Interventional Strategies
Brief Title: Understanding Local Determinants of Cardiovascular Disease and Diabetes
Status: Completed | Type: Observational
Sponsor: Malawi Epidemiology and Intervention Research Unit (Other)
Responsible Party: Sponsor
Other Study IDs: NCD
Record Dates: First submitted 2018-01-30; First posted 2018-02-05 (Actual); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Hypertension; Diabetes; Overweight and Obesity
MeSH Terms: conditions — Hypertension; Diabetes Mellitus; Overweight; Obesity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Cross-sectional survey of all adults residing in two defined geographical regions in urban Lilongwe and rural Karonga District. Participants were interviewed, had anthropometric measures taken, and had fasting blood specimens taken.

ELIGIBILITY:
Inclusion Criteria:

* all adults over 18 self-identifying as normally resident in the pre-defined geographical areas

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All adults within 2 defined geographical areas - one in urban Lilongwe, one in rural Karonga District
Sampling Method: Probability Sample
Enrollment: 28891 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
What is the true burden of hypertension, diabetes, and hyperlipidaemia? | By end of 2018
  Prevalence of hypertension (BP <140/90 or self-report of antihypertensive use), diabetes (fasting blood glucose >7.0 or self-report history of diabetes), and hyperlipidaemia

SECONDARY OUTCOMES:
What is the prevalence of known risk factors - notably smoking, obesity, physical inactivity, alcohol, salt, and saturated fat intake? | By end of 2020
  Description of prevalence of known risk factors of hypertension, diabetes, and hyperlipidaemia.
  Dietary salt intake is estimated both by how long a defined quantity of salt is reported to last in a household on average, and from spot urine sodium specimens.
Is infection, notably HIV infection or its therapy, associated with increased risk of NCDs? | By end of 2020
  Description of HIV infection and its therapy in relationship to hypertension, diabetes and hyperlipidaemia

CONTACTS AND LOCATIONS:
Locations (1):
- MEIRU, Lilongwe, Malawi

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Prynn JE, Banda L, Amberbir A, Price AJ, Kayuni N, Jaffar S, Crampin AC, Smeeth L, Nyirenda M. Dietary sodium intake in urban and rural Malawi, and directions for future interventions. Am J Clin Nutr. 2018 Sep 1;108(3):587-593. doi: 10.1093/ajcn/nqy125. PMID 29982267